CLINICAL TRIAL: NCT01325389
Title: Effects of Myo-inositol Plus Melatonin in Perimenopausal Women
Brief Title: Myo-inositol Plus Melatonin in Perimenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Myo+MEL_peri_women
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Perimenopause

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myo+Mel (Experimental): Patients are treated with 2g of myo + 3mg of melatonin daily
  Interventions: Dietary Supplement: Myo-Mel
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Myo-Mel
  Arms: Myo+Mel
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Menopause is the milestone of a more broaden condition that can last up to 10 years. The first menopausal symptoms usually appear around the age of 42 and are characterized by a gradual decline in thyroid and gonadal function with a progressive increase of plasmatic luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels.

Recent studies have shown that myo-inositol and melatonin play a major role in ovarian homeostasis. In particular, it has been demonstrated that myo-inositol and/or melatonin supplementation lead to an increase of oocyte quality.

Additional studies focused on postmenopausal women have shown that myo-inositol is able to ameliorate the metabolic syndrome that often affects these patients, thus reducing the risk of cardiovascular diseases (CVDs).

The aim of the present study is to evaluate whether myo-inositol and melatonin might play a positive role in regulating hormonal levels during menopausal onset.

ELIGIBILITY:
Inclusion Criteria:

* FSH between 15 and 50 IU/ml on the 5th day of the menses
* Oligomenorrhea

Exclusion Criteria:

-

Ages: 42 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- AGUNCO, Rome, Italy

REFERENCES:
- [Background] Papaleo E, Unfer V, Baillargeon JP, Fusi F, Occhi F, De Santis L. RETRACTED: Myo-inositol may improve oocyte quality in intracytoplasmic sperm injection cycles. A prospective, controlled, randomized trial. Fertil Steril. 2009 May;91(5):1750-1754. doi: 10.1016/j.fertnstert.2008.01.088. Epub 2008 May 7. PMID 18462730
- [Background] Rizzo P, Raffone E, Benedetto V. Effect of the treatment with myo-inositol plus folic acid plus melatonin in comparison with a treatment with myo-inositol plus folic acid on oocyte quality and pregnancy outcome in IVF cycles. A prospective, clinical trial. Eur Rev Med Pharmacol Sci. 2010 Jun;14(6):555-61. PMID 20712264
- [Background] Giordano D, Corrado F, Santamaria A, Quattrone S, Pintaudi B, Di Benedetto A, D'Anna R. Effects of myo-inositol supplementation in postmenopausal women with metabolic syndrome: a perspective, randomized, placebo-controlled study. Menopause. 2011 Jan;18(1):102-4. doi: 10.1097/gme.0b013e3181e8e1b1. PMID 20811299
- [Background] Tamura H, Nakamura Y, Korkmaz A, Manchester LC, Tan DX, Sugino N, Reiter RJ. Melatonin and the ovary: physiological and pathophysiological implications. Fertil Steril. 2009 Jul;92(1):328-43. doi: 10.1016/j.fertnstert.2008.05.016. Epub 2008 Sep 18. PMID 18804205
- [Background] Tamura H, Takasaki A, Miwa I, Taniguchi K, Maekawa R, Asada H, Taketani T, Matsuoka A, Yamagata Y, Shimamura K, Morioka H, Ishikawa H, Reiter RJ, Sugino N. Oxidative stress impairs oocyte quality and melatonin protects oocytes from free radical damage and improves fertilization rate. J Pineal Res. 2008 Apr;44(3):280-7. doi: 10.1111/j.1600-079X.2007.00524.x. PMID 18339123